CLINICAL TRIAL: NCT06157281
Title: Combining Positive Deviance and Implementation Science to Improve Retention in HIV Care in South Africa
Brief Title: Positive Deviance to Improve Retention in HIV Care HIV Care in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Stellenbosch (Other); Western Cape Department of Health and Wellness (Unknown)
Responsible Party: Principal Investigator, Allison Ober, Senior Health Policy Researcher, RAND
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HCAAD058-1000; R34MH119889 (NIH)
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: 3 lower-retention clinics will receive the intervention. Outcomes will be compared to those at all other lower-retention clinics of the same type within the same health system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect Intervention (Experimental): HIV providers withing each clinic will participate in the Intervention. The intervention, called "Connect," consists of several strategies within three domains, as follows:
  Domain 1: Engage, Encourage, Support Staff
  Strategy 1a: Monthly staff huddle with staff recognition activities and compassion-focused rounds
  Strategy 1b: Compassion training
  Domain 2: Create a welcome physical environment
  Strategy 2a: Aesthetic improvements toward a warm, welcoming environment
  Domain 3: Expedite and workflow practices
  Strategy 3a: Pre-pull patient folders; hold folders for immediate tracking; map patients to identify locations
  Strategy 3b: Integrate welcome-back services for those who miss follow-up appointments
  Interventions: Behavioral: Connect
- Control (No Intervention): Staff in control clinics will not receive an intervention.

INTERVENTIONS:
Behavioral: Connect — A multicomponent, clinic-level intervention consisting of strategies aimed at improving retention and viral load suppression by enhancing the patient and staff experience.
  Arms: Connect Intervention

SUMMARY:
The goal of this pilot trial is to test the effectiveness of a newly developed multicomponent clinic-level intervention for improving retention in HIV care among people living with HIV in South Africa. The intervention was developed based on intensive study of clinics with high retention rates. The main question this study aims to answer is: Does the intervention improve retention in HIV care for people with HIV (PWH)?

The intervention, called "Connect," consists of several strategies within three domains, as follows:

Domain 1: Engage, Encourage, Support Staff

Strategy 1a: Monthly staff huddle with staff recognition activities and compassion-focused rounds

Strategy 1b: Compassion training

Domain 2: Create a welcome physical environment

Strategy 2a: Aesthetic improvements toward a warm, welcoming environment

Domain 3: Expedite and augment workflow practices

Strategy 3a: Pre-pull patient folders; hold folders for immediate tracking; map patients to identify locations

Strategy 3b: Integrate welcome-back services for those who miss follow-up appointments

HIV staff at three clinics with below-average retention rates who consent to participate will take part in intervention activities. Results will be compared to those of all other lower-retention clinics within the same health system.

DETAILED DESCRIPTION:
The goal of this pilot trial is to test the effectiveness of a newly developed multicomponent clinic-level intervention for improving retention in HIV care among people living with HIV in South Africa. The intervention is based on intensive interviews, focus groups and surveys conducted with HIV staff within 3 clinics in a health system with lower-than-average retention rates. The next step is to conduct a pilot trial to test whether the intervention can improve care for people living with HIV.

The main question this study aims to answer is: Does the intervention improve retention in HIV care for people with HIV (PWH)?

The intervention, called "Connect," consists of several strategies within three domains, as follows:

Domain 1: Engage, Encourage, Support Staff

Strategy 1a: Monthly staff huddle with staff recognition activities and compassion-focused rounds. Each clinic holds a monthly huddle toward team cohesion, support and a shared vision for retention. Consists of some core activities, such as "Rounds", staff recognition; and activities to build team cohesion and staff wellbeing.

Strategy 1b: Compassion training. Based on evidenced-based compassion training, train and support staff on interacting with other providers and patients in compassionate ways.

Domain 2: Create a welcome physical environment.

Strategy 2a: Aesthetic improvements toward a warm, welcoming environment. Examples include bright paint in waiting areas, murals on outside walls, plants, posters with positive messaging on walls.

Domain 3: Expedite and augment workflow practices.

Strategy 3a: Pre-pull patient folders; hold folders for immediate tracking; map patients to identify locations. Staff pull folders for next-day appointments, communicate no-shows with trackers, use mapping to have patients indicate approximate living areas to facilitate tracking.

Strategy 3b: Welcome-back services for those who miss follow-up appointments. Integrate specialized, patient-centered services for those who miss their 1-month or 3-month visit to re-enter care easily. The key elements of this are genuine concern for the patient, avoiding scolding or blaming the patients, checks on patient health and symptoms, and exploration of barriers including how to overcome these and facilitate ongoing treatment.

HIV staff at three clinics with below-average retention rates who consent to participate will take part in intervention activities. Results will be compared to those of all other lower-retention clinics within the same health system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Administrator or other staff member of one of three participating clinics

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Antiretroviral Therapy (ART) Retention | 6 months
  Proportion of patients in care at the same clinic 6 months after ART initiation
Viral Load Suppression (VLS) | 6 months
  Proportion of patients with VLS 6 months* after initiating ART (<50 copies/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Allison J Ober, PhD, Principal Investigator — RAND
Locations (1):
- Western Cape Department of Health and Wellbeing CDH or CHC, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
Aggregated retention and VLS data by clinic can be made available to other researchers.